CLINICAL TRIAL: NCT00274196
Title: A Prospective Study of the Specificity and Sensitivity of Ultrasound in Diagnosing Occult Hip Fractures
Brief Title: Ultrasound as a Diagnostic Tool for Occult Hip Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 28-17.02.06-HMO-CTIL
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2007-11-14 (Estimated); Status verified 2007-11

CONDITIONS: Occult Fractures
Keywords: fractures, occult; hip; ultrasound examination; MRI; sensitivity; specificity
MeSH Terms: conditions — Fractures, Closed; Hypersensitivity | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: ultrasound examination — a single time 10 minutes procedure within the first week after the injury
Procedure: MRI scan — a single time 30 minutes procedure, performed always after the ultrasound scan

SUMMARY:
The purpose of this study is to measure the sensitivity and specificity of ultrasound exam of the hip in diagnosing occult hip fractures.

DETAILED DESCRIPTION:
Introduction: Most hip fractures are diagnosed by history, physical examination and confirmed by plain radiographs. When initial X-rays are negative or equivocal, and there is a clinical suspicion of occult hip fracture, additional diagnostic tests are necessary such as MRI which is expensive and in many hospitals less available, or bone scan which needs to be delayed 48-72 hours from injury to be indicative. Ultrasound examination has been shown to be an accurate measurement to diagnose occult fractures in the ankle and is a relatively easy, available, non-expansive examination. We propose the use of bedside ultrasound examination of the hip as a screening tool for occult hip fractures.

Objective: To measure the sensitivity and specificity of ultrasound exam of the hip in diagnosing or ruling out occult hip fractures.

Materials and methods: We will include all patients 40 years and older with a painful hip after an injury, and with "normal" hip X-rays. Each patient will undergo two hip ultrasounds by two different examiners. Afterwards, the patients will undergo MRI of the hip. The MRI will serve as the gold standard for treatment decisions. The results of the ultrasound will be compared to the MRI to evaluate its sensitivity and specificity.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 years or older, with suspected hip fracture but normal plain X-rays

Exclusion Criteria:

* Patients younger than 40 years and with contra-indications for MRI scan

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-02; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Comparison between ultrasound exam and MRI (sensitivity and specificity) | 2008

CONTACTS AND LOCATIONS:
Overall Officials: Ori Safran, MD, Principal Investigator — Hadassah Medical Organization; Charles Milgrom, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Lubovsky O, Liebergall M, Mattan Y, Weil Y, Mosheiff R. Early diagnosis of occult hip fractures MRI versus CT scan. Injury. 2005 Jun;36(6):788-92. doi: 10.1016/j.injury.2005.01.024. Epub 2005 Apr 7. PMID 15910835